CLINICAL TRIAL: NCT00511459
Title: A Randomized, 4-Arm, Placebo-Controlled Phase 2 Trial of AMG 386 in Combination With Bevacizumab and Paclitaxel or AMG 386 Plus Paclitaxel as First-Line Therapy in Subjects With Her2-Negative, Metastatic or Locally Recurrent Breast Cancer
Brief Title: Phase 2 Study of AMG 386 Plus Paclitaxel With or Without Bevacizumab as First Line Therapy in Her2-Negative Breast Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20060341
Record Dates: First submitted 2007-08-02; First posted 2007-08-03 (Estimated); Last update posted 2015-10-29 (Estimated); Status verified 2015-10

CONDITIONS: Locally Recurrent and Metastatic Breast Cancer
Keywords: Randomized; 4-Arm; Placebo controlled; Phase 2 Trial; AMG 386; Paclitaxel; Bevacizumab; First-line Therapy; Her-2 Negative; Metastatic or Locally Recurrent Breast Cancer
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — trebananib; Bevacizumab; Paclitaxel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- A (Experimental): Paclitaxel 90 mg/m² IV QW (3 on/1 off) + bevacizumab 10 mg/kg IV Q2W + AMG 386 10 mg/kg IV QW
  Interventions: Drug: Bevacizumab; Drug: AMG 386; Drug: Paclitaxel
- D (Experimental): Paclitaxel 90 mg/m² IV QW (3 on/1 off) + Open Label AMG 386 10 mg/kg IV QW
  Interventions: Drug: AMG 386; Drug: Paclitaxel
- B (Experimental): Paclitaxel 90 mg/m² IV QW (3 on/1 off) + bevacizumab 10 mg/kg IV Q2W + AMG 386 3 mg/kg IV QW
  Interventions: Drug: AMG 386; Drug: Bevacizumab; Drug: Paclitaxel
- C (Active Comparator): Paclitaxel 90 mg/m² IV QW (3 on/1 off) + bevacizumab 10 mg/kg IV Q2W + AMG 386 placebo IV QW
  Interventions: Drug: AMG 386 Placebo; Drug: Bevacizumab; Drug: Paclitaxel

INTERVENTIONS:
Drug: AMG 386 Placebo — AMG 386 Placebo [blinded]
  Arms: C
Drug: AMG 386 — AMG 386 3mg/kg IV QW [blinded]
  Arms: B
Drug: Bevacizumab — Bevacizumab 10mg/kg IV Q2W
  Arms: A; B; C
Drug: AMG 386 — AMG 386 10mg/kg IV QW [Open-Label]
  Arms: D
Drug: AMG 386 — AMG 386 10mg/kg IV QW [blinded]
  Arms: A
Drug: Paclitaxel — Paclitaxel 90mg/m2 IV QW (3 on/1 0ff)

SUMMARY:
This is a phase 2, randomized, placebo controlled, multi-center study to estimate the treatment effect and evaluate the safety and tolerability of AMG 386 in combination with paclitaxel and paclitaxel/bevacizumab in the treatment of subjects with Her2-negative metastatic or locally recurrent breast cancer.

AMG 386 is a man-made medication that is designed to stop the development of blood vessels in cancer tissues. Cancer tissues rely on the development of new blood vessels, a process called angiogenesis, to obtain a supply of oxygen and nutrients to grow.

DETAILED DESCRIPTION:
Primary Objective: To estimate the treatment effect as measured by progression free survival (PFS) of subjects receiving AMG 386 (at 2 doses) in combination with paclitaxel + bevacizumab relative to paclitaxel + bevacizumab + placebo.

Secondary Objective(s):

* To compare the treatment effect as measured by PFS of subjects receiving open-label AMG 386 in combination with paclitaxel relative to paclitaxel + bevacizumab + placebo
* To compare the treatment effect as measured by PFS of subjects receiving AMG 386 in combination with paclitaxel and bevacizumab relative to paclitaxel + AMG 386
* To evaluate the safety and tolerability of the combination and non-bevacizumab regimens
* To estimate other measures (RR, DOR, TTR, TTP) of treatment effect
* To evaluate the pharmacokinetics (PK) of AMG 386 and bevacizumab when used in combination
* To estimate the incidence of anti-AMG386 antibody formation

Exploratory Objective(s):

* To explore the pharmacodynamic (PD) response as assessed by changes in blood levels of angiogenic cytokines, tumor apoptosis, and other markers
* To explore the association of histological features and selected immunologic, biochemical, pharmacogenetic, or angiogenic markers in tumor biopsies, plasma, or serum samples with safety and/or efficacy outcomes

Study Design:

This is a phase 2, randomized, placebo controlled, multi-center study to estimate the treatment effect and evaluate the safety and tolerability of AMG 386 in combination with paclitaxel and paclitaxel/bevacizumab in the treatment of subjects with Her2-negative metastatic or locally recurrent breast cancer.

Two hundred twenty subjects will be randomized 1:1:1:1 to each of the following arms:

Arm A: Paclitaxel 90 mg/m² IV QW (3 on/1 off) + bevacizumab 10 mg/kg IV Q2W + AMG 386 10 mg/kg IV QW Arm B: Paclitaxel 90 mg/m² IV QW (3 on/1 off) + bevacizumab 10 mg/kg IV Q2W + AMG 386 3 mg/kg IV QW Arm C: Paclitaxel 90 mg/m² IV QW (3 on/1 off) + bevacizumab 10 mg/kg IV Q2W + AMG 386 placebo IV QW Arm D: Paclitaxel 90 mg/m² IV QW (3 on/1 off) + Open Label AMG 386 10 mg/kg IV QW To maintain the double-blind in arms A, B, and C, each subject will be infused weekly with a volume of investigational product equivalent to 10 mg/kg AMG 386 IV. Arm D will receive open label AMG 386 and will not receive a placebo for bevacizumab.

Subjects will be discontinued from study treatment at any time for radiographic disease progression, clinical progression, unacceptable toxicity, subject withdrawal of consent, or death.

Subjects alive at the time of discontinuation of all study medications will be followed for up to 48 months from the date of the last subject enrolled into the trial to evaluate overall survival.

Radiological imaging to assess disease status will be performed every 8 weeks ± 7 days (2 cycles) for 2 years and then every 4 months ± 1 month thereafter during the study until subjects develop radiographic disease progression per the modified RECIST criteria. In addition, any subject who discontinues study drug treatment prior to disease progression will continue to have radiological imaging performed every 8 weeks ± 7 days during the long term follow up period if the subject has not been in the study for 2 years until the subject develops radiographic disease progression or begins a new treatment. If the subject has been on study for 2 years, radiological imaging every 4 months ± 1 month will be performed during long term follow-up period until the subject develops radiographic disease progression or begins a new treatment.

The overall study design is described by a study schema immediately following this synopsis. Amgen Global Safety (AGS) will charter a data review team (DRT) that is independent of the team conducting the study and will review unblinded safety data after 20, 40, and 80 subjects have been randomized and have had the opportunity to receive at least 1 cycle (4 weeks) of study treatment.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have histologically or cytologically confirmed adenocarcinoma of the breast with locally recurrent or metastatic disease. Locally recurrent disease must not be amenable to resection with curative intent.
* Measurable or non-measurable disease per modified RECIST guidelines
* ECOG of 0 or 1 (within 14 days prior to randomization)
* Adequate organ and hematological function as evidenced by the following laboratory studies within 14 days prior to randomization:

  • Cardiac function, as follows:
* Normal sinus rhythm (no significant ECG changes)
* Left ventricular ejection fraction ≥ LLN, as determined by echocardiogram or MUGA scan, according to institutional standards within 28 days prior to randomization

Exclusion Criteria:

* Inflammatory Breast Cancer
* Common Terminology Criteria for Adverse Events (CTCAE) Version 3.0 peripheral neuropathy > grade 1 at randomization
* History of arterial or venous thrombosis, including transient ischemic attack (TIA), within 1 year prior to randomization
* Adjuvant or neoadjuvant taxane treatment within 12 months of randomization. Any other adjuvant chemotherapy regimen must be discontinued at least 21 days prior to randomization
* Prior chemotherapy, vaccine, or biological therapy for locally recurrent or metastatic breast cancer (prior endocrine therapy is permitted)
* Prior radiation therapy, radiofrequency ablation, percutaneous cryotherapy or hepatic chemoembolization on all sites of disease unless disease progression was subsequently documented 14 days prior to randomization.
* Overexpression of HER-2 (gene amplification by FISH or 3+ over expression by immunohistochemistry).
* Current or prior history of central nervous system metastasis
* History of bleeding diathesis or clinically significant bleeding within 6 months prior to randomization
* Major surgical procedure within 28 days prior to randomization
* Open breast biopsy within 14 days prior to randomization
* Minor surgical procedure, placement of access device, or fine needle aspiration within 7 days of first dose
* Prior malignancy (other than thyroid cancer, in situ cervical cancer, or basal cell cancer of the skin, treated with curative intent and without evidence of disease for ≥ 3 years prior to randomization)
* Clinically significant cardiac disease within 12 months prior to randomization, including myocardial infarction, unstable angina, grade 2 or greater peripheral vascular disease, cerebrovascular accident, transient ischemic attack, congestive heart failure, or arrhythmias not controlled by outpatient medication
* Non-healing wound, ulcer or fracture
* Known hypersensitivity to paclitaxel or drugs using the vehicle cremophor
* Known hypersensitivity to bacterial proteins, or any of the drugs required in this study
* Known positive test for human immunodeficiency virus (HIV), hepatitis C, or hepatitis B surface antigen
* Known active or chronic hepatitis
* Uncontrolled hypertension as defined as systolic blood pressure ≥ 150 mm Hg and diastolic blood pressure ≥ 90 mm Hg. Anti-hypertensive medications are allowed if the subject is stable on their current dose at the time of randomization
* Currently or previously treated with any VEGF or VEGFr inhibitor, including but not limited to, bevacizumab, SU11248 (sunitinib), PTK787 (vatalinib), AZD 2171, AEE-788, BAY 43-9006 (sorafenib) and AMG 706.
* Treatment with coumarin-type anticoagulants, (other than low dose prophylaxis for central venous catheters ≤ 1mg/day) within 7 days prior to randomization
* Currently or previously treated with angiopoietin inhibitors, or inhibitors of TIE-1 or TIE-2 including, but not limited to, AMG 386, XL880, XL820
* Treatment with immune modulators such as cyclosporine and tacrolimus within 30 days prior to randomization
* Concomitant therapy with any hormonal agent such as raloxifene, tamoxifen, or other selective estrogen receptor modulators (SERMS), given for breast cancer prevention or for osteoporosis. Subjects must have discontinued these agents 28 days prior to randomization
* Pregnant (ie, positive beta-human chorionic gonadotropin test) or is breast feeding

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 228 (Actual)
Dates: Start 2007-07; Primary Completion 2010-08 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | 3 YEARS

SECONDARY OUTCOMES:
Objective Response (OR) | 3 YEARS
Duration of Response (DOR) | 3 YEARS
Time to response | 3 YEARS
Overall Survival | 3 YEARS
Time to progression (TTP) | 3 YEARS
Incidence of AEs and significant laboratory changes | 3 YEARS
AMG 386 Pharmakokinetic parameters | 3 YEARS
Incidence of the occurrence of anti-AMG 386 antibody formation | 3 YEARS

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (73):
- United States (26):
  - Research Site, Litchfield Park, Arizona
  - Research Site, Tucson, Arizona
  - Research Site, Hot Springs, Arkansas
  - Research Site, Little Rock, Arkansas
  - Research Site, Campbell, California
  - Research Site, Los Angeles, California
  - Research Site, Murrieta, California
  - Research Site, Santa Maria, California
  - Research Site, New Haven, Connecticut
  - Research Site, Stamford, Connecticut
  - Research Site, Orlando, Florida
  - Research Site, Robbinsdale, Minnesota
  - Research Site, Henderson, Nevada
  - Research Site, Lebanon, New Hampshire
  - Research Site, Nashua, New Hampshire
  - Research Site, Edison, New Jersey
  - Research Site, Mountain Lakes, New Jersey
  - Research Site, Asheville, North Carolina
  - Research Site, Charlotte, North Carolina
  - Research Site, Hershey, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Columbia, South Carolina
  - Research Site, Richardson, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Sugar Land, Texas
  - Research Site, Ogden, Utah
- Australia (6):
  - Research Site, Kurralta Park, South Australia
  - Research Site, Epping, Victoria
  - Research Site, Fitzroy, Victoria
  - Research Site, Footscray, Victoria
  - Research Site, Malvern, Victoria
  - Research Site, Perth, Western Australia
- Austria (3):
  - Research Site, Innsbruck
  - Research Site, Vienna
  - Research Site, Wels
- Belgium (3):
  - Research Site, Leuven
  - Research Site, Liège
  - Research Site, Wilrijk
- Research Site, Herlev, Denmark
- Research Site, Helsinki, Finland
- France (7):
  - Research Site, La Roche-sur-Yon
  - Research Site, Lyon
  - Research Site, Marseille
  - Research Site, Montpellier
  - Research Site, Paris
  - Research Site, Toulouse
  - Research Site, Vandœuvre-lès-Nancy
- Hungary (4):
  - Research Site, Gyula
  - Research Site, Kaposvár
  - Research Site, Szombathely
  - Research Site, Veszprém
- India (6):
  - Research Site, Bangalore, Karnataka
  - Research Site, Miraj, Maharashtra
  - Research Site, Mumbai, Maharashtra
  - Research Site, Nagpur, Maharashtra
  - Research Site, Pune, Maharashtra
  - Research Site, Jaipur, Rajasthan
- Research Site, Maastricht, Netherlands
- Poland (5):
  - Research Site, Gdansk
  - Research Site, Lubin
  - Research Site, Poznan
  - Research Site, Warsaw
  - Research Site, Wroclaw
- Spain (4):
  - Research Site, JaÃ©n, AndalucÃ-a
  - Research Site, Sabadell, CataluÃ±a
  - Research Site, Santiago de Compostela, Galicia
  - Research Site, Madrid, Madrid
- United Kingdom (6):
  - Research Site, Guildford
  - Research Site, Leicester
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Northwood
  - Research Site, Nottingham

REFERENCES:
- [Derived] Dieras V, Wildiers H, Jassem J, Dirix LY, Guastalla JP, Bono P, Hurvitz SA, Goncalves A, Romieu G, Limentani SA, Jerusalem G, Lakshmaiah KC, Roche H, Sanchez-Rovira P, Pienkowski T, Segui Palmer MA, Li A, Sun YN, Pickett CA, Slamon DJ. Trebananib (AMG 386) plus weekly paclitaxel with or without bevacizumab as first-line therapy for HER2-negative locally recurrent or metastatic breast cancer: A phase 2 randomized study. Breast. 2015 Jun;24(3):182-90. doi: 10.1016/j.breast.2014.11.003. Epub 2015 Mar 5. PMID 25747197
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com